CLINICAL TRIAL: NCT00481793
Title: Germline Genetic Variation and Risk of Chromosome Aberrations Among Mayak Nuclear Workers
Brief Title: Relationship of Genetic Differences to the Development of Chromosome Abnormalities
Status: Terminated | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999904215; 04-C-N215; NCT00342901 (obsolete NCT alias); NCT01338168 (obsolete NCT alias)
Record Dates: First submitted 2007-06-01; First posted 2007-06-04 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-09-17

CONDITIONS: Radiation Exposure
Keywords: Plutonium; Ionizing Radiation; Polymorphism; Biological Marker; Russia

SUMMARY:
This is a collaborative study by the National Cancer Institute, Columbia University, and the Southern Urals Biophysics Institute in Russia. It will examine the relationship of differences in certain genes to the development of chromosomal abnormalities in workers at the Mayak nuclear production plant in Ozyorsk, Russia. This population was exposed to higher radiation doses from external and internal sources than those received by their counterparts in other countries or considered permissible today. If a risk relationship is found between genetic differences and chromosome abnormalities, the information might be useful in studies designed to examine how high radiation exposures cause cancer.

Radiation-exposed Mayak workers employed from 1948 to 1972 in the three Ozyorsk plants directly related to nuclear weapons production may be eligible for this study. They must have remained local residents in the area and estimates of their external and internal radiation exposures must be available.

Participants provide a blood sample for genetic studies and answer a questionnaire that includes demographic information and information about their family health history, history of benign tumors, if any, and history of smoking and alcohol consumption. Additional information is collected from patients' medical records.

...

DETAILED DESCRIPTION:
Greater understanding of the role of individual variation in response to radiation exposure might clarify the inconsistent relationship between radiation dose, intermediate markers of induced DNA damage, and subsequent cancer risk. REB proposes to collaborate with Columbia University and the Southern Urals Biophysics Institute to elucidate the contribution of germline genetic variation to the frequency of chromosomal aberrations in a cohort of Russian nuclear workers with notable and atypical radiation exposures. Our collaborators are utilizing a new biodosimetry method, termed mBAND, to measure intra-chromosomal aberrations, a potentially useful biomarker of exposure to high linear energy transfer radiation such as plutonium. In addition, they will assess inter-chromosomal aberrations using mFISH (multicolor fluorescent insitu hybridization). As factors other than radiation dose may influence aberration frequency, REB proposes to add to this DOE-funded study an investigation of germline genetic variation in DNA repair and other genes in relation to aberration risk. Mayak nuclear workers (n = approximately 350) employed from 1948-72 will receive a short questionnaire and have a blood sample drawn while receiving routine annual medical exams. Germline genotype will be assessed as a risk factor for chromosome aberration frequency. In this study, we have the opportunity to address scientific questions regarding radiation carcinogenesis mechanisms at relatively little cost in a population with rare, higher dose exposures.

ELIGIBILITY:
* INCLUSION CRITERIA - EXPOSED POPULATION:

Individuals eligible to be included in the 'exposed' population include all those employed from 1948-1972 in the three plants directly related to nuclear-weapon production (nuclear reactor, radiochemical production plant, plutonium production plant), who have remained local residents, and who have estimates of their external gamma dose and internal plutonium exposure.

Some eligible workers did not have any plutonium exposure, but are still eligible to be included in the exposed sample due to their external radiation exposure.

All participants are required to be cancer-free at the time of enrollment.

EXCLUSION CRITERIA - EXPOSED POPULATION:

Individuals who have a medical history of radiation therapy or a blood transfusion within the previous year will be excluded.

As the sample size would not be adequate to examine their risk separately, Tartars and Bashkirs will not be included in the study.

INCLUSION CRITERIA - COMPARISON GROUP:

The comparison population will be drawn from current and former workers in the auxiliary plants (water treatment facility and mechanical repair plant) at the Mayak facility.

Included will be a stratified random sample of these workers who were employed from 1948-1972, who have remained local residents, and who have estimates of their external gamma dose.

Individuals selected will be frequency-matched according to age (5 year age groups) and gender to the exposed worker population.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2004-06-09; Study Completion 2014-09-17

CONTACTS AND LOCATIONS:
Overall Officials: Martha Linet, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Southern Urals Biophysics Institute, Ozersk, Russia

REFERENCES:
- [Background] Bonassi S, Hagmar L, Stromberg U, Montagud AH, Tinnerberg H, Forni A, Heikkila P, Wanders S, Wilhardt P, Hansteen IL, Knudsen LE, Norppa H. Chromosomal aberrations in lymphocytes predict human cancer independently of exposure to carcinogens. European Study Group on Cytogenetic Biomarkers and Health. Cancer Res. 2000 Mar 15;60(6):1619-25. PMID 10749131
- [Background] Cardis E, Gilbert ES, Carpenter L, Howe G, Kato I, Armstrong BK, Beral V, Cowper G, Douglas A, Fix J, et al. Effects of low doses and low dose rates of external ionizing radiation: cancer mortality among nuclear industry workers in three countries. Radiat Res. 1995 May;142(2):117-32. PMID 7724726
- [Background] Dupont WD, Plummer WD Jr. Power and sample size calculations for studies involving linear regression. Control Clin Trials. 1998 Dec;19(6):589-601. doi: 10.1016/s0197-2456(98)00037-3. PMID 9875838